CLINICAL TRIAL: NCT01304654
Title: Practice of Mechanical Ventilation in Pediatric Oncologic Patients Diagnosed with Acute Lung Injury / Acute Respiratory Distress Syndrome
Brief Title: ALI (Acute Lung Injury) /ARDS (Acute Respiratory Distress Syndrome) in Oncologic Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, Rodrigo Genaro Arduini, MD, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Other Study IDs: UTI/IOP 02/11; 0031/11 (Other: CEP UNIFESP)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2013-03

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Neoplasms
Keywords: acute lung injury; respiratory distress syndrome; neoplasms; child
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALI/ARDS oncologic patients: Consecutively admitted patients at GRAACC's PICU with malignancy diagnosis according to IDC-10, in a 24mo consecutive period, under mechanical ventilation for over 24h and with ALI/ARDS criteria, not younger than 29 days or older than 17 years 11 months

SUMMARY:
Identify pediatric oncologic patients with ALI/ARDS at GRAACC (Grupo de Apoio ao Adolescente e a Criança com Câncer) /IOP's (Instituto de Oncologia Pediátrica) Pediatric Intensive Care Unit and evaluate the mechanical ventilation practice in these subjects for a 48mo period.

DETAILED DESCRIPTION:
Evaluate adequate mechanical ventilation based on protective ventilation protocols for children available so far.

Evaluate and describe the subjects. Evaluate the necessity and outcome of rescue therapies (surfactant, prone position, corticosteroids, alveolar recruitment) Obtain data about ALI/ARDS' etiology, mortality rates and predictive factors related to the outcomes (PICU/ hospital discharge or death)

ELIGIBILITY:
Inclusion Criteria:

* patients admitted at the intensive care unit with diagnosis of acute lung injury or acute respiratory distress syndrome and submitted to mechanical ventilation for over 24h

Exclusion Criteria:

* mechanical ventilation less than 24h
* absence of ALI/ARDS criteria
* no neoplasm diagnosis

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric oncologic patients
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-01-08; Primary Completion 2013-03-30 (Actual); Study Completion 2013-06-15 (Actual)

PRIMARY OUTCOMES:
Identify pediatric oncologic patients with ALI/ARDS at GRAACC's PICU and evaluate how they are mechanically ventilated | 2y

SECONDARY OUTCOMES:
Epidemiologic data about the selected patients | 28 days
  Type and data about their mechanical ventilation, etiologic factors for ALI/ARDS, mortality rates, predictive factors about outcomes (death/ discharge), necessity and types of rescue therapies (surfactant, prone position, corticosteroids, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo G Arduini, MD, Principal Investigator — Grupo de Apoio ao Adolescente e a Crianca com Cancer
Locations (1):
- Grupo de Apoio ao Adolescente e à Criança com Câncer, São Paulo, São Paulo, Brazil